CLINICAL TRIAL: NCT01549652
Title: 5HT3 Antagonists to Treat Opioid Withdrawal and to Prevent the Progression of Physical Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Larry Fu-nien Chu, Principle Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 5HT3 19821; 1R01DA029078 (NIH)
Record Dates: First submitted 2012-02-13; First posted 2012-03-09 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Opioid Withdrawal; Physical Dependence
MeSH Terms: interventions — Ondansetron; Morphine; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevention of Opioid Withdrawal (Experimental): Chronic back pain patients will titrate onto sustained release oral morphine for 30 days, and then will be randomized to take either ondansetron 8 mg or matching placebo thirty minutes prior to naloxone-induced withdrawal in clinic (Naloxone 0.4 mg/70 kg; if deemed necessary by the clinician to induce withdrawal, a second naloxone dose may be administered at 0.8 mg/70 kg). Participants will return to their titrated morphine dose for one week and then return for the opposite pre-treatment followed by naloxone-induced withdrawal in clinic. Participants will then taper back to their original dose of morphine for one week.
  Interventions: Drug: Ondansetron; Drug: Placebo; Drug: Morphine; Drug: Naloxone 0.4 mg/70 kg; Drug: Naloxone 0.8 mg/70 kg
- Prevention of Physical Dependence (Experimental): Chronic back pain patients will titrate onto sustained release oral morphine for 30 days; during morphine treatment, participants will be randomized to take either ondansetron 8 mg or matching placebo three times daily along with the oral morphine treatment. After thirty days, participants will return to the lab to undergo naloxone-induced withdrawal in clinic (Naloxone 0.4 mg/70 kg; if deemed necessary by the clinician to induce withdrawal, a second naloxone dose may be administered at 0.8 mg/70 kg). Participants will then taper back to their original dose of morphine for one week.
  Interventions: Drug: Ondansetron; Drug: Placebo; Drug: Morphine; Drug: Naloxone 0.4 mg/70 kg; Drug: Naloxone 0.8 mg/70 kg

INTERVENTIONS:
Drug: Ondansetron — Ondansetron 8 mg oral tablet
  Other Names: Zofran
Drug: Placebo — Placebo to Match Ondansetron
Drug: Morphine — Sustained release oral morphine, beginning at 30 mg/d, titrated up by 15 mg/d every 2 days until adequate analgesia is achieved
Drug: Naloxone 0.4 mg/70 kg — Naloxone 0.4 mg/70 kg intravenous
Drug: Naloxone 0.8 mg/70 kg — Naloxone 0.8 mg/70 kg intravenous

SUMMARY:
Opioid medications are commonly used for pain relief. When given over time, physical dependence can occur. This results in unpleasant side effects (such as agitation and nausea) if opioid medications are suddenly stopped. This study aims to test the use of the drug ondansetron to reduce the symptoms associated with opioid withdrawal and to prevent the progression of opioid physical dependence, thereby allowing future investigators to better test the role of physical dependence in the development of addiction and also possibly improving acceptance of abstinence-based programs for addiction.

DETAILED DESCRIPTION:
This study will be split into two separate investigations, aim 1 and aim 2.

Study aim 1 (Prevention of Opioid Withdrawal) will investigate whether ondansetron, a 5HT3-receptor antagonist, can reduce or prevent withdrawal signs and symptoms in patients physically dependent on opioids to treat chronic back pain. In this aim, study participants will be titrated onto sustained release oral morphine for 30 days after which time they will return to the lab to undergo naloxone-induced withdrawal with either 8 mg ondansetron pre-treatment (30 min prior to naloxone-induced withdrawal) or placebo. Participants will then return to their titrated dose of oral morphine for one week before returning for the second study session in which they will receive the opposite pre-treatment (8 mg ondansetron or placebo) 30 minutes prior to naloxone-induced withdrawal. Objective opioid withdrawal score (OOWS), subjective opioid withdrawal score (SOWS) and Profile of Mood States (POMS) will be assessed at baseline and five or seven times during the study sessions at 30 and 37 days post titration. Beck Depression Inventory, Roland-Morris Questionnaire and State-Trait Anxiety Inventory and VAS Pain Score will be assessed at baseline as well as at both study sessions (30 and 37 days post titration).

Study aim 2 (Prevention of Physical Dependence) will investigate whether ondansetron, a 5HT3 receptor antagonist, can prevent physical dependence in patients taking opioids chronically for controlling chronic back pain. Participants will taper onto sustained release oral morphine for 10 days then will maintain the effective dose for twenty days (total of 30 days) while simultaneously taking 8 mg ondansetron or placebo three times daily with morphine dose. After 30 days of morphine plus 8 mg ondansetron or placebo, study participants will return to the lab to undergo naloxone-induced withdrawal. OOWS, SOWS, POMS, pain visual analogue scale (VAS), Beck Depression Inventory and Roland Morris Disability Index will be administered at baseline and at the beginning of each study session (30 days post titration). Furthermore OOWS, SOWS and POMS will be administered twice during the first study session and at least five times during the second study session (Day 30): at the beginning of the session, after IV insertion, and after naloxone-induced opioid withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic low-back pain and who may be taking up to 30 mg equivalent of morphine per day (such as Vicodin, Percocet, etc)
* 18-60 years old
* Eligible to escalate opioid therapy dose, as determined by the treating physician or PI
* At low risk for addiction as determined by the PI and an addiction expert, Dr. Ian Carroll.

Exclusion Criteria:

* History of cardiovascular disease
* History of peripheral neuropathic pain, scleroderma, or other condition that would preclude cold water forearm immersion
* History of addiction or chronic pain conditions other than low-back pain, d) history of cardiac arrhythmia
* History of hepatic disease
* Use of steroid or nerve-stimulating medications
* Any condition precluding opioid use
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry F Chu, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu LF, Liang DY, Li X, Sahbaie P, D'arcy N, Liao G, Peltz G, David Clark J. From mouse to man: the 5-HT3 receptor modulates physical dependence on opioid narcotics. Pharmacogenet Genomics. 2009 Mar;19(3):193-205. doi: 10.1097/FPC.0b013e328322e73d. PMID 19214139
- [Background] Atlas SJ, Nardin RA. Evaluation and treatment of low back pain: an evidence-based approach to clinical care. Muscle Nerve. 2003 Mar;27(3):265-84. doi: 10.1002/mus.10311. PMID 12635113
- [Background] Betses M, Brennan T. Abusive prescribing of controlled substances--a pharmacy view. N Engl J Med. 2013 Sep 12;369(11):989-91. doi: 10.1056/NEJMp1308222. Epub 2013 Aug 21. No abstract available. PMID 23964897
- [Background] Birnbaum HG, White AG, Schiller M, Waldman T, Cleveland JM, Roland CL. Societal costs of prescription opioid abuse, dependence, and misuse in the United States. Pain Med. 2011 Apr;12(4):657-67. doi: 10.1111/j.1526-4637.2011.01075.x. Epub 2011 Mar 10. PMID 21392250
- [Background] Chu LF, D'Arcy N, Brady C, Zamora AK, Young CA, Kim JE, Clemenson AM, Angst MS, Clark DJ. Analgesic tolerance without demonstrable opioid-induced hyperalgesia: a double-blinded, randomized, placebo-controlled trial of sustained-release morphine for treatment of chronic nonradicular low-back pain. Pain. 2012 Aug;153(8):1583-1592. doi: 10.1016/j.pain.2012.02.028. Epub 2012 Jun 16. PMID 22704854
- [Background] Clark JD. Chronic pain prevalence and analgesic prescribing in a general medical population. J Pain Symptom Manage. 2002 Feb;23(2):131-7. doi: 10.1016/s0885-3924(01)00396-7. PMID 11844633
- [Background] Colthup PV, Felgate CC, Palmer JL, Scully NL. Determination of ondansetron in plasma and its pharmacokinetics in the young and elderly. J Pharm Sci. 1991 Sep;80(9):868-71. doi: 10.1002/jps.2600800913. PMID 1839313
- [Background] Compton P, Athanasos P, Elashoff D. Withdrawal hyperalgesia after acute opioid physical dependence in nonaddicted humans: a preliminary study. J Pain. 2003 Nov;4(9):511-9. doi: 10.1016/j.jpain.2003.08.003. PMID 14636819
- [Background] Compton P, Miotto K, Elashoff D. Precipitated opioid withdrawal across acute physical dependence induction methods. Pharmacol Biochem Behav. 2004 Feb;77(2):263-8. doi: 10.1016/j.pbb.2003.10.017. PMID 14751453
- [Background] Handelsman L, Cochrane KJ, Aronson MJ, Ness R, Rubinstein KJ, Kanof PD. Two new rating scales for opiate withdrawal. Am J Drug Alcohol Abuse. 1987;13(3):293-308. doi: 10.3109/00952998709001515. PMID 3687892
- [Background] Plosker GL, Milne RJ. Ondansetron: a pharmacoeconomic and quality-of-life evaluation of its antiemetic activity in patients receiving cancer chemotherapy. Pharmacoeconomics. 1992 Oct;2(4):285-304. doi: 10.2165/00019053-199202040-00005. PMID 10147044
- [Background] Meert TF. Effects of various serotonergic agents on alcohol intake and alcohol preference in Wistar rats selected at two different levels of alcohol preference. Alcohol Alcohol. 1993 Mar;28(2):157-70. PMID 8517886
- [Result] Chu LF, Sun J, Clemenson A, Erlendson MJ, Rico T, Cornell E, Obasi H, Sayyid ZN, Encisco EM, Yu J, Gamble JG, Carroll I, Clark JD. Ondansetron Does Not Reduce Withdrawal in Patients With Physical Dependence on Chronic Opioid Therapy. J Addict Med. 2017 Sep/Oct;11(5):342-349. doi: 10.1097/ADM.0000000000000321. PMID 28514235
- [Result] Chu LF, Rico T, Cornell E, Obasi H, Encisco EM, Vertelney H, Gamble JG, Crawford CW, Sun J, Clemenson A, Erlendson MJ, Okada R, Carroll I, Clark JD. Ondansetron does not prevent physical dependence in patients taking opioid medications chronically for pain control. Drug Alcohol Depend. 2018 Feb 1;183:176-183. doi: 10.1016/j.drugalcdep.2017.06.043. Epub 2017 Aug 14. PMID 29278818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chronic back pain patients were recruited from the San Francisco Bay Area via recruitment posters, newspaper advertisements, and radio and television announcements.
Pre-assignment Details: No enrolled participants were excluded from the study after enrollment and before assignment to groups.
Groups:
- Prevention of Opioid Withdrawal-Ondansetron; Prevention of Opioid Withdrawal-Placebo: Chronic back pain patients titrated onto sustained release oral morphine for 30 days, then were randomized to take either ondansetron 8 mg or matching placebo thirty minutes prior to naloxone-induced withdrawal in clinic (naloxone dose: 0.4 mg/70 kg; if deemed necessary by the clinician to induce withdrawal, a second naloxone dose may be administered at 0.8 mg/70 kg). Participants returned to their titrated morphine dose for one week and then returned for the opposite pre-treatment followed by naloxone-induced withdrawal in clinic. Participants then tapered back to their original dose of morphine for one week.
  Data regarding how many participants received ondansetron first versus placebo first are not accessible.
- Prevention of Physical Dependence - Ondansetron; Prevention of Physical Dependence - Placebo: Chronic back pain patients titrated onto sustained release oral morphine for 30 days; during morphine treatment, participants were randomized to take either ondansetron 8 mg or matching placebo three times daily along with the oral morphine treatment. After thirty days, participants returned to the lab to undergo naloxone-induced withdrawal in clinic (naloxone dose: 0.4 mg/70 kg; if deemed necessary by the clinician to induce withdrawal, a second naloxone dose may have been administered at 0.8 mg/70 kg). Participants then tapered back to their original dose of morphine for one week.
Period: Overall Study
Arm/Group | Prevention of Opioid Withdrawal-Ondansetron | Prevention of Opioid Withdrawal-Placebo | Prevention of Physical Dependence - Ondansetron | Prevention of Physical Dependence - Placebo
Started | 27 | 30 | 40 | 36
Completed | 15 | 18 | 23 | 25
Not Completed | 12 | 12 | 17 | 11
Not completed — Did Not Receive Allocated Intervention | 0 | 0 | 2 | 0
Not completed — Study Drug Titration Failure | 5 | 6 | 0 | 0
Not completed — Withdrawal Effect | 0 | 2 | 0 | 0
Not completed — Did Not Return Due to Withdrawal Effect | 5 | 1 | 0 | 0
Not completed — Problem with Infusion | 1 | 0 | 0 | 0
Not completed — Titration Non-Compliance | 1 | 3 | 4 | 5
Not completed — Titration Side Effects | 0 | 0 | 6 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Participants that completed the protocol are included in the analysis
Groups:
- Prevention of Opioid Withdrawal: Chronic back pain patients titrated onto sustained release oral morphine for 30 days, then were randomized to take either ondansetron 8 mg or matching placebo thirty minutes prior to naloxone-induced withdrawal in clinic (naloxone dose: 0.4 mg/70 kg; if deemed necessary by the clinician to induce withdrawal, a second naloxone dose may be administered at 0.8 mg/70 kg). Participants returned to their titrated morphine dose for one week and then returned for the opposite pre-treatment followed by naloxone-induced withdrawal in clinic. Participants then tapered back to their original dose of morphine for one week.
  Data regarding how many participants received ondansetron first versus placebo first are not accessible.
- Prevention of Physical Dependence-Ondansetron; Prevention of Physical Dependence-Placebo: Chronic back pain patients titrated onto sustained release oral morphine for 30 days; during morphine treatment, participants were randomized to take either ondansetron 8 mg or matching placebo three times daily along with the oral morphine treatment. After thirty days, participants returned to the lab to undergo naloxone-induced withdrawal in clinic (naloxone dose: 0.4 mg/70 kg; if deemed necessary by the clinician to induce withdrawal, a second naloxone dose may have been administered at 0.8 mg/70 kg). Participants then tapered back to their original dose of morphine for one week.
- Total: Total of all reporting groups
Arm/Group | Prevention of Opioid Withdrawal | Prevention of Physical Dependence-Ondansetron | Prevention of Physical Dependence-Placebo | Total
Number analyzed (Participants) | 33 | 23 | 25 | 81
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 33 | 23 | 25 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 12 | 35
  Male | 20 | 13 | 13 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Objective Opioid Withdrawal Score (OOWS) From Baseline (Prevention of Opioid Withdrawal)
Description: Originally developed by Handelsman, the Objective Opioid Withdrawal Scale (OOWS) score is a well-characterized measure of opioid withdrawal in humans, calculated as the sum of a 13-item physician assessment documenting physically observable signs of withdrawal, which are rated as present (1) or absent (0) during the observation period. The minimum score of 0 means the patient is not showing any signs of opioid withdrawal. The maximum score of 13 signifies all signs of opioid withdrawal to the largest extent possible.
  Immediately prior to ondansetron or placebo administration a baseline OOWS score was taken. 30 minutes later participants received naloxone, then 15 minutes later an OOWS score was taken. If deemed necessary by the clinician, participants may have received a second naloxone dose (25 minutes following 1st naloxone dose), then 15 minutes later an OOWS score was taken. Change from the baseline OOWS score to the score assessed following the last naloxone dose is reported.
Time Frame: Baseline; 15 minutes following last naloxone dose
Population: Participants in the Prevention of Opioid Withdrawal Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prevention of Opioid Withdrawal: Chronic back pain patients titrated onto sustained release oral morphine for 30 days, then were randomized to take either ondansetron 8 mg or matching placebo thirty minutes prior to naloxone-induced withdrawal in clinic (naloxone dose: 0.4 mg/70 kg; if deemed necessary by the clinician to induce withdrawal, a second naloxone dose may be administered at 0.8 mg/70 kg). Participants returned to their titrated morphine dose for one week and then returned for the opposite pre-treatment followed by naloxone-induced withdrawal in clinic. Participants then tapered back to their original dose of morphine for one week.
Arm/Group | Prevention of Opioid Withdrawal
Number analyzed (Participants) | 33
units on a scale
  Change in OOWS (Ondansetron) | 3.6 (2.2)
  Change in OOWS (Placebo) | 3.6 (2.4)
Statistical Analysis 1: Comparison: Prevention of Opioid Withdrawal; For the purposes of our post-hoc power calculation we considered a 30% treatment effect clinically significant. Based on the mean observed OOWS score during withdrawal during the placebo session and the variance of that mean score and assuming a paired data analysis and an alpha of 0.05, we found that we had 80% power to detect a treatment effect as low as 25% reduction in OOWS; Test type: Superiority or Other; p = 0.87, t-test, 2 sided — Students' t-tests for paired samples with Bonferroni correction for multiple comparisons were used to compare differences between the outcome measures for crossover treatment arms (placebo vs. ondansetron)

2. Secondary Outcome: Change in Subjective Opioid Withdrawal Score (SOWS) From Baseline (Prevention of Opioid Withdrawal)
Description: The Subjective Opioid Withdrawal Score (SOWS) score is calculated as the sum of 16 subjective patient-reported symptom scores rated on a scale of 0 to 4 (0=not at all, 4=extremely) based on what subjects were experiencing at the time of testing. A maximum score of 64 would suggest the patient is experiencing the symptoms of withdrawal to the maximum extent possible while the lowest score of 0 would suggest the patient is not experiencing any of the symptoms of withdrawal. Immediately prior to ondansetron or placebo administration a baseline SOWS score was taken. 30 minutes later participants received naloxone, then 15 minutes later an SOWS score was taken. If necessary (as deemed by the clinician), participants may have received a second naloxone dose (25 minutes following 1st naloxone dose), then 15 minutes later an SOWS score was taken. Change from the baseline SOWS score to the score assessed following the last naloxone dose is reported
Time Frame: Baseline; 15 minutes following last naloxone dose
Population: Participants in the Prevention of Opioid Withdrawal Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Opioid Withdrawal
Number analyzed (Participants) | 33
units on a scale
  Change in SOWS (Ondansetron) | 12.5 (11.2)
  Change in SOWS (Placebo) | 12.2 (10.7)
Statistical Analysis 1: Comparison: Prevention of Opioid Withdrawal; Test type: Superiority or Other; p = 0.92, t-test, 2 sided

3. Secondary Outcome: Beck Depression Inventory Score (BDIS) Change From Baseline (Prevention of Opioid Withdrawal)
Description: The Beck Depression Inventory (a 21-item self-report multiple-choice inventory) yields a single summed score between 0 and 63; higher scores indicate more severe depression. Change is from baseline score (taken at the beginning of the first study visit, prior to beginning of titration into morphine) to the score taken after taking morphine for 30 days (score taken prior to receiving ondansetron or placebo, at the beginning of second study visit).
Time Frame: 2 study days 1 month apart (at the start of each study visit)
Population: Participants in the Prevention of Opioid Withdrawal Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Opioid Withdrawal
Number analyzed (Participants) | 33
units on a scale | -0.44 (3.36)
Statistical Analysis 1: Comparison: Prevention of Opioid Withdrawal; Test type: Superiority or Other; p = 0.47, t-test, 2 sided

4. Secondary Outcome: Profile of Mood States (POMS) Change in Score From Baseline (Prevention of Opioid Withdrawal)
Description: Profile of Mood States (POMS) is a 65-question survey of how participants have been feeling over the past week, assessing tension, depression, anger, fatigue, confusion and vigor. Each question is on a 5-point scale: 0 (not at all) to 4 (extremely). Overall score range: 0 to 200 (lower scores corresponding to fewer symptoms), calculated by adding total scores for tension, depression, anger, fatigue and confusing, and subtracting that total score from the total score for vigor. Immediately prior to ondansetron or placebo administration a baseline POMS score was taken. 30 minutes later participants received naloxone, then 15 minutes later a POMS score was taken. If necessary (as deemed by the clinician), participants may have received a second naloxone dose (25 minutes following 1st naloxone dose), then 15 minutes later an POMS score was taken. Change from the baseline POMS score to the score assessed following the last naloxone dose is reported.
Time Frame: Baseline; 15 minutes following last naloxone dose
Population: Participants in the Prevention of Opioid Withdrawal Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Opioid Withdrawal
Number analyzed (Participants) | 33
units on a scale
  Change in POMS Score (Ondansetron) | 29.3 (31.3)
  Change in POMS Score (Placebo) | 28.3 (37.1)
Statistical Analysis 1: Comparison: Prevention of Opioid Withdrawal; Test type: Superiority or Other; p = 0.91, t-test, 2 sided

5. Secondary Outcome: Change in Pain Visual Analog Scale (VAS) From Baseline (Prevention of Opioid Withdrawal)
Description: The VAS is a 0 to 100 millimeter scale where 0 corresponds to no pain and 100 to extreme pain, used by participants to indicated their level of pain over the last two weeks. Change is from baseline score for average level of pain (taken at the beginning of the first study visit, prior to beginning of titration into morphine) to the score taken after taking morphine for 30 days (score taken prior to receiving ondansetron or placebo, at the beginning of second study visit).
Time Frame: 2 study days 1 month apart (at the start of each study visit)
Population: Participants in the Prevention of Opioid Withdrawal Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Opioid Withdrawal
Number analyzed (Participants) | 33
units on a scale | -2.68 (2.23)
Statistical Analysis 1: Comparison: Prevention of Opioid Withdrawal; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Change in Roland-Morris Disability Index (RMDI) From Baseline (Prevention of Opioid Withdrawal)
Description: The Roland-Morris Disability Index is a 24-question instrument used to assess level of disability from lower back pain. Scores range from 0-24 with lower scores corresponding to fewer symptoms. Change is from baseline score (taken at the beginning of the first study visit, prior to beginning of titration into morphine) to the score taken after taking morphine for 30 days (score taken prior to receiving ondansetron or placebo, at the beginning of second study visit).
Time Frame: 2 study days 1 month apart (at the start of each study visit)
Population: Participants in the Prevention of Opioid Withdrawal Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Opioid Withdrawal
Number analyzed (Participants) | 33
units on a scale | -2.59 (4.56)
Statistical Analysis 1: Comparison: Prevention of Opioid Withdrawal; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

7. Primary Outcome: Change in Objective Opioid Withdrawal Score From Baseline (Prevention of Physical Dependence)
Description: Originally developed by Handelsman, the OOWS score is a well-characterized measure of opioid withdrawal in humans, calculated as the sum of a 13-item physician assessment documenting physically observable signs of withdrawal, which are rated as present (1) or absent (0) during the observation period. The maximum score is 13 and suggests the patient is showing all signs of opioid withdrawal to the largest extent possible. The minimum score of 0 suggests the patient is not showing any signs of opioid withdrawal.
  Immediately prior to ondansetron or placebo administration a baseline OOWS score was taken. 30 minutes later participants received naloxone, then 15 minutes later an OOWS score was taken. If necessary (as deemed by the clinician), participants may have received a second naloxone dose (25 minutes following 1st naloxone dose), then 15 minutes later an OOWS score was taken. Change from the baseline OOWS score to the score assessed following the last naloxone dose is reported.
Time Frame: Baseline; 15 minutes following last naloxone dose
Population: Participants in the Prevention of Physical Dependence Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prevention of Physical Dependence: Chronic back pain patients titrated onto sustained release oral morphine for 30 days; during morphine treatment, participants were randomized to take either ondansetron 8 mg or matching placebo three times daily along with the oral morphine treatment. After thirty days, participants returned to the lab to undergo naloxone-induced withdrawal in clinic (naloxone dose: 0.4 mg/70 kg; if deemed necessary by the clinician to induce withdrawal, a second naloxone dose may have been administered at 0.8 mg/70 kg). Participants then tapered back to their original dose of morphine for one week.
Arm/Group | Prevention of Physical Dependence
Number analyzed (Participants) | 48
units on a scale
  Change in OOWS (Ondansetron): number analyzed (Participants) | 23
  Change in OOWS (Ondansetron) | 4.5 (2.5)
  Change in OOWS (Placebo): number analyzed (Participants) | 25
  Change in OOWS (Placebo) | 4.2 (2.4)
Statistical Analysis 1: Comparison: Prevention of Physical Dependence; We aimed for a 20% change in OOWS score to show the treatment effect with a power of 80% and an alpha of 0.05, yielding a target of 23 patients per treatment group; Test type: Superiority or Other; p = 0.6, t-test, 2 sided — Students' t-test for paired samples were used to compare differences between the outcome measures for treatment groups (placebo vs. ondansetron)

8. Secondary Outcome: Change in Subjective Opioid Withdrawal Score From Baseline (Prevention of Physical Dependence)
Description: The SOWS score is composed of 16 subjective symptoms rated on a scale of 0 to 4 (0=not at all, 4=extremely) based on what subjects were experiencing at the time of testing. A maximum score of 64 would suggest the patient is experiencing the symptoms of withdrawal to the maximum extent possible while the lowest score of 0 would suggest the patient is not experiencing any of the symptoms of withdrawal. Immediately prior to ondansetron or placebo administration a baseline SOWS score was taken. 30 minutes later participants received naloxone, then 15 minutes later an SOWS score was taken. If necessary (as deemed by the clinician), participants may have received a second naloxone dose (25 minutes following 1st naloxone dose), then 15 minutes later an SOWS score was taken. Change from the baseline SOWS score to the score assessed following the last naloxone dose is reported
Time Frame: Baseline; 15 minutes following last naloxone dose
Population: Participants in the Prevention of Physical Dependence Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Physical Dependence
Number analyzed (Participants) | 48
units on a scale
  Change in SOWS (Ondansetron): number analyzed (Participants) | 23
  Change in SOWS (Ondansetron) | 16.4 (13.1)
  Change in SOWS (Placebo): number analyzed (Participants) | 25
  Change in SOWS (Placebo) | 12.0 (10.0)
Statistical Analysis 1: Comparison: Prevention of Physical Dependence; Test type: Superiority or Other; p = 0.20, t-test, 2 sided

9. Secondary Outcome: Beck Depression Inventory Score (BDIS) Change From Baseline (Prevention of Physical Dependence)
Description: The Beck Depression Inventory (a 21-item self-report multiple-choice inventory) yields a single summed score between 0 and 63; higher scores indicate more severe depression. Change is from baseline score (taken at the beginning of the first study visit, prior to beginning of titration into morphine) to the score taken after taking morphine for 30 days (score taken at the beginning of second study visit).
Time Frame: 2 study days 1 month apart (at the start of each study visit)
Population: Participants in the Prevention of Physical Dependence Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Physical Dependence
Number analyzed (Participants) | 48
units on a scale
  Change in BDIS (Ondansetron): number analyzed (Participants) | 23
  Change in BDIS (Ondansetron) | -0.6 (2.6)
  Change in BDIS (Placebo): number analyzed (Participants) | 25
  Change in BDIS (Placebo) | 0.2 (3.1)
Statistical Analysis 1: Comparison: Prevention of Physical Dependence; Test type: Superiority or Other; p = 0.34, t-test, 2 sided

10. Secondary Outcome: Profile of Mood States (POMS) Change in Score From Baseline (Prevention of Physical Dependence)
Description: (Profile of Mood States) POMS is a 65-question survey of how participants have been feeling over the past week, assessing tension, depression, anger, fatigue, confusion and vigor. Each question is on a 5-point scale: 0 (not at all) to 4 (extremely). Overall score range: 0 to 200 (lower scores corresponding to fewer symptoms), calculated by adding total scores for tension, depression, anger, fatigue and confusing, and subtracting that total score from the total score for vigor. Immediately prior to ondansetron or placebo administration a baseline POMS score was taken. 30 minutes later participants received naloxone, then 15 minutes later a POMS score was taken. If necessary (as deemed by the clinician), participants may have received a second naloxone dose (25 minutes following 1st naloxone dose), then 15 minutes later an POMS score was taken. Change from the baseline POMS score to the score assessed following the last naloxone dose is reported.
Time Frame: Baseline; 15 minutes following last naloxone dose
Population: Participants in the Prevention of Physical Dependence Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Physical Dependence
Number analyzed (Participants) | 48
units on a scale
  Change in POMS (Ondansetron): number analyzed (Participants) | 23
  Change in POMS (Ondansetron) | 36.1 (27.6)
  Change in POMS (Placebo): number analyzed (Participants) | 25
  Change in POMS (Placebo) | 29.2 (26.3)
Statistical Analysis 1: Comparison: Prevention of Physical Dependence; Test type: Superiority or Other; p = 0.40, t-test, 2 sided

11. Secondary Outcome: Change in Pain Visual Analog Scale (VAS) From Baseline (Prevention of Physical Dependence)
Description: The VAS is a 0 to 100 millimeter scale where 0 corresponds to no pain and 100 to extreme pain, used by participants to indicated their level of pain over the last two weeks. Change is from baseline score for average level of pain (taken at the beginning of the first study visit, prior to beginning of titration into morphine) to the score taken after taking morphine for 30 days (score taken at the beginning of second study visit).
Time Frame: 2 study days 1 month apart (at the start of each study visit)
Population: Participants in the Prevention of Physical Dependence Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Physical Dependence
Number analyzed (Participants) | 48
units on a scale
  Change in VAS Score (Ondansetron): number analyzed (Participants) | 23
  Change in VAS Score (Ondansetron) | -2.9 (1.4)
  Change in VAS Score (Placebo): number analyzed (Participants) | 25
  Change in VAS Score (Placebo) | -2.8 (1.9)
Statistical Analysis 1: Comparison: Prevention of Physical Dependence; Test type: Superiority or Other; p = 0.84, t-test, 2 sided

12. Secondary Outcome: Change in Roland-Morris Disability (RMDI) Index From Baseline (Prevention of Physical Dependence)
Description: The Roland-Morris Disability Index is a 24-question instrument used to assess level of disability from lower back pain. Scores range from 0-24 with lower scores corresponding to fewer symptoms. Change is from baseline score (taken at the beginning of the first study visit, prior to beginning of titration into morphine) to the score taken after taking morphine for 30 days (score taken at the beginning of second study visit).
Time Frame: 2 study days 1 month apart (at the start of each study visit)
Population: Participants in the Prevention of Physical Dependence Arm were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevention of Physical Dependence
Number analyzed (Participants) | 48
units on a scale
  Change in RMDI (Ondansetron): number analyzed (Participants) | 23
  Change in RMDI (Ondansetron) | -4.6 (4.2)
  Change in RMDI (Placebo): number analyzed (Participants) | 25
  Change in RMDI (Placebo) | -2.0 (3.1)
Statistical Analysis 1: Comparison: Prevention of Physical Dependence; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Prevention of Opioid Withdrawal | Prevention of Physical Dependence
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/48
Other Adverse Events (participants affected / at risk) | 0/33 | 0/48

LIMITATIONS AND CAVEATS:
Aim 1: Use of a single 8mg dose of ondansetron as well as a lack of biochemical data is a limitation of this study.

Aim 2: Use of 8mg of ondansetron instead of varying doses is a limitation of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes